CLINICAL TRIAL: NCT00005423
Title: Dietary Quality and Subsequent Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4341; R03HL048530 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2002-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To examine dietary quality and subsequent cardiovascular disease (CVD).

DETAILED DESCRIPTION:
BACKGROUND:

Although considerable evidence exists for associations between diet and subsequent cardiovascular disease (CVD) among younger and middle-aged adults, no comprehensive studies of these relationships have been conducted using a national sample of older Americans. National guidelines have recommended reductions of dietary fat, saturated fat, cholesterol and sodium as dietary practice to reduce CVD. However, it is possible that the focus on eliminating dietary components may obscure the advantages of consuming diets that are nutritionally adequate.

Findings from this study could have important implications for setting research priorities to further study the effects of specific dietary variables on CVD, and for implementing national nutrition policies to assist Americans in selecting healthy diets.

DESIGN NARRATIVE:

Data from NHANES I and the three cycles of NHANES I Epidemiologic Followup Study (NHEFS) were used to 1) to examine the associations between several measures of dietary quality at baseline and subsequent 14-year morbidity and mortality from CVD for a national sample of 6109 United States adults aged 45 to 74 years at baseline; 2) to assess the relative importance of the associations of dietary quality and CVD for older adults compared to middle-aged adults. Dietary variables were based on responses to the 24-hour dietary recall and the food frequency questionnaire administered at baseline and included a composite measure of dietary quality, intakes of specific nutrients, and usual consumption of foods from 19 food groups. Baseline measures used as covariates included body mass index, blood pressure, serum cholesterol, sociodemographic variables (e.g., age, race, income, occupation), behavioral variables (e.g., smoking, alcohol consumption, activity level), and chronic health conditions. CVD outcomes were determined from medical history questionnaires, hospital records and death certificates. Change in blood pressure between baseline and 10-year followup were examined as an outcome variable as well as a covariate in the association between diet and CVD.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1992-07; Study Completion 1994-12 (Actual)